CLINICAL TRIAL: NCT01864928
Title: Reperfusion in Acute Stroke - Creating the Clinical Decision-Making Tool (RESOLVE)
Brief Title: Rapid Evaluation for Stroke Outcomes Using Lytics in Vascular Event (RESOLVE) Registry and Implementation Quality Improvement Study
Acronym: RESOLVE
Status: Completed | Type: Observational
Sponsor: Saint Luke's Health System (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28677
Record Dates: First submitted 2013-05-14; First posted 2013-05-30 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic stroke; ePRISM
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stroke population: Adults with ischemic stroke.

SUMMARY:
Despite abundant evident supporting the use of acute reperfusion therapy in the setting of acute ischemic stroke (AIS), adoption of this practice in routine clinical care is poor. We hypothesize that a significant barrier is the difficulty in weighing the benefits and risks of rt-PA treatment in the care of an individual patient, a problem compounded by the time urgency of decision-making and clinical fears that weigh risks of treatment more heavily than benefits.

The goal of this Quality Improvement (QI) study is to leverage an IT solution that we have developed, ePRISM, that executes multivariable risk models with patient-specific data so that a personalized estimate of an individual's outcomes (both risks and benefits) with and without rt-PA, can be generated so support safer, more effective clinical care. Through an earlier project, we will have programmed ePRISM with the best available risk-stratification models and developed a clinically useful format for presenting the data to support clinical decision-making in AIS.

Through QI, we propose to identify the optimal mechanism for integrating the tool within the routine flow of patient care in preparation for more definitive studies, or dissemination strategies, to improve the treatment of patients with AIS.

DETAILED DESCRIPTION:
Specific Aim 1: Implement ePRISM and the RESOLVE Decision Aid (DA) at 2 sites (Saint Luke's Hospital in Kansas City and Saint Luke's North) for Emergency Department (ED) access and decision support.

1. Procedures and Evaluation

1. Map process flow and define the optimal points of care for both the informed consent and decision aid.
2. Pre-implementation registry or data retrieval of patient/family satisfaction with information during consent process pre-PRISM, as well as time from presentation to treatment.
3. Implementation of ePRISM software and the RESOLVE DA.
4. Monitor proportion of patients in whom the RESOLVE DA is used.
5. Post-implementation registry or data retrieval of patient/family satisfaction and knowledge, as well as time from presentation to treatment.
6. Interviews of providers on confidence in making treatment decisions.
7. Monitor patient outcomes through 90 day follow up phone call as per the standard of care.

Specific Aim 2: Implement ePRISM and the RESOLVE DA onsite at the the Barnes Jewish Hospital Emergency Department. After optimizing the integration of ePRISM and the RESOLVE DA at Saint Luke's Hospital and Saint Luke's North, we will evaluate strategies for implementation at Barnes Jewish Hospital's Emergency Department Telestroke Program.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* 18 years of age or older

Exclusion Criteria:

* Active internal bleeding
* History of cerebrovascular accident
* Evidence of intracranial hemorrhage on pretreatment evaluation
* Suspicion of subarachnoid hemorrhage on pretreatment evaluation
* Recent (within 3 months) intracranial or intraspinal surgery, serious head trauma, or previous stroke
* History of intracranial hemorrhage
* Uncontrolled hypertension at time of treatment
* Seizure at the onset of stroke
* Intracranial neoplasm, arteriovenous malformation, or aneurysm
* Known bleeding diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Successful implementation of ePRISM and the RESOLVE DA in 3 ED's and a telestroke program. | 2 years
  Successful implementation of ePRISM and the RESOLVE DA in 3 ED's and a telestroke program. Successful implementation is defined as: 1) the activation of ePRISM and generation the RESOLVE DA by ePRISM; 2) the staff and clinician's reported value of the new RESOLVE DA for use during the rt-PA decision making process.

SECONDARY OUTCOMES:
Patient/family satisfaction. | 2 years
  Patient/family satisfaction with PRISM for Acute Ischemic Stroke (AIS).
Knowledge transfer. | 2 years
  Knowledge transfer of AIS and rt-PA risks and benefits through survey.

CONTACTS AND LOCATIONS:
Overall Officials: John A Spertus, MD, MPH, Principal Investigator — St. Luke's Hospital, Kansas City, Missouri; Carole Decker, MSN, PhD, Study Director — St. Luke's Hospital, Kansas City, Missouri

REFERENCES:
- [Derived] Decker C, Chhatriwalla E, Gialde E, Garavalia B, Summers D, Quinlan ME, Cheng E, Rymer M, Saver JL, Chen E, Kent DM, Spertus JA. Patient-Centered Decision Support in Acute Ischemic Stroke: Qualitative Study of Patients' and Providers' Perspectives. Circ Cardiovasc Qual Outcomes. 2015 Oct;8(6 Suppl 3):S109-16. doi: 10.1161/CIRCOUTCOMES.115.002003. PMID 26515198